CLINICAL TRIAL: NCT03257319
Title: Inhaled Versus Intravenous Opioid Dosing for the Initial Treatment of Severe Acute Pain in the Emergency Department
Brief Title: Inhaled vs IV Opioid Dosing for the Initial Treatment of Severe Acute Pain in the Emergency Department
Acronym: CLIN-AEROMORPH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014/0009/HP
Record Dates: First submitted 2017-07-20; First posted 2017-08-22 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Pain, Acute; Emergencies; Morphine
MeSH Terms: conditions — Acute Pain; Emergencies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- inhaled morphine + IV placebo (Experimental): Arm A: inhaled titration of morphine chlorhydrate+ IV placebo
  Interventions: Drug: inhaled titration of morphine chlorhydrate; Drug: IV placebo
- IV morphine +inhaled placebo (Placebo Comparator): Arm B:IV titration of morphine chlorhydrate + inhaled placebo
  Interventions: Device: Inhaled placebo; Drug: IV titration of morphine chlorhydrate

INTERVENTIONS:
Drug: inhaled titration of morphine chlorhydrate — Patient in arm A will receive 1 to 3 titration
  Other Names: IV placebo
  Arms: inhaled morphine + IV placebo
Drug: IV placebo — Patient in arm A will receive 1 to 6 injection
  Other Names: inhaled titration of morphine chlorhydrate
  Arms: inhaled morphine + IV placebo
Device: Inhaled placebo — Patient in arm B will receive 1 to 3 titration
  Other Names: IV titration of morphine chlorhydrate
  Arms: IV morphine +inhaled placebo
Drug: IV titration of morphine chlorhydrate — Patient in arm BA will receive 1 to 6 injection
  Other Names: Inhaled placebo
  Arms: IV morphine +inhaled placebo

SUMMARY:
Prospective single-blind, multicenter, national, randomized, controlled trial in 15 Emergency Department to compare two ways of morphine titration. The eligible patient is included immediately after his arrival in the Emergency Department, after being questioned by the triage nurse about the presence and the intensity of pain, when the VAS is greater than 70 (or EN>7) and after written consent.

After installation into the examination room, patient is randomized in one of two parallel groups (stratified by sex and center using software) and receives one of the two treatments, either inhaled morphine + IV placebo or IV morphine+ inhaled placebo (control group).

In both groups, titration is defined by a dose of repeated boluses as long as the relief is not achieved (VAS> 30 or EN >3) and the criteria to stop titration are not met.

A 5 minutes time interval between the boluses is chosen. Each aerosol takes 5 minutes at a constant air flow, aerosol mask, plastic tubing and PVC transparent tank are used.

Thus patient receives a maximum of 3 aerosol (one aerosol every 10 minutes) and a maximum of 6 IV injections (one injection every 5 minutes) The stopping criteria, except pain relief, are linked to the occurrence of side effects and specific cares are described into the protocol (in case of severe ventilatory depression naloxone titration is provided). Exit criteria from the emergency room and from the hospital are defined. An information sheet is delivered.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and <75 years old;
* EVA ≥ 70/100 or EN ≥ 7/10;
* Patient who received clear information from the investigator and read and signed the consent form;
* Patient affiliated with, or beneficiary of a social security category;
* For women:

O of childbearing age: effective contraception (oral contraception, intrauterine device or use of condoms) O menopausal status (amenorrhoea less than 12 months before the inclusion visit) O objectivized sterility (diagnosis or surgically)

Exclusion Criteria:

* Chronic pain (> 3 months)
* Taking opioids longer than 10 days (including "weak" opioids tramadol and / or codeine);
* Taking Rifampicin;
* Impaired ability to discern, cognitive impairment;
* Morphine-related contraindications:

O Obstructive chronic obstructive or restrictive respiratory failure known or suspected compensated or not, O Hypersensitivity to the active substance or to any of the excipients, O Severe hepatocellular insufficiency (known or suspected), O Chronic renal failure known or suspected, O Uncontrolled epilepsy, O Cranial trauma (intracranial hypertension), O Associations with buprenorphine, nalbuphine, pentazocine and naltrexone

* Active drug history or practice (s);
* Evidence of reduced fracture or dislocation in emergency rooms;
* Suspected occlusive syndrome
* SaO2 <95%;
* FR <12 / min;
* Glasgow <15 or other alertness disorders;
* HR heart rate <50 bpm and / or Auriculo-Ventricular block (PR XML File Identifier: zR6XOYKSEQ9GjQHghP8c465EwF0= Page 15/30 interval> 200 ms);
* Arterial hypotension with systolic blood pressure TA syst <100 mm Hg;
* Pregnant or nursing
* Persons deprived of their liberty by an administrative or judicial decision, a person placed under the safeguard of justice, guardianship;
* Patients with poor comprehension of spoken or written French;
* Patients participating in another interventional clinical study;
* Contra-indication related to the use of saline solution
* Contra-indications related to the use of aerosol:

O Necessity to access the face O Allergy known to plastic

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Rate of relief obtained or "success rate" at 1 hour from the start of drug administration, and not at the end of titration, such as EVA1 ≤ 30/100 (or EN1 ≤ 3/10). | 1 hour after the initiation of the titration
  Rate of relief obtained or "success rate" at 1 hour from the start of drug administration, and not at the end of titration, such as EVA1 ≤ 30/100 (or EN1 ≤ 3/10).

SECONDARY OUTCOMES:
Evaluate antalgic efficacy criteria | From the beginning of the titration until the end of the titration- assessed within one day
  Quantity of morphine administered from the beginning of the titration until the end of the titration
Evaluate antalgic efficacy criteria | From the beginning of the titration until the end of the titration- assessed up to one day
  Delay between first administration of Morphine and EVA ≤ 30 or EN ≤ 3 obtained
Evaluate antalgic efficacy criteria | From the beginning of the titration until the end of the titration- assessed up to one day
  Delay between first administration of Morphine and EVA ≤ 30 or EN ≤ 3 obtained for patient treated only with morphine IV
Evaluate antalgic efficacy criteria | From the beginning of the titration until the end of the titration- assessed up to one day
  Number of patients with EVA ≤ 30 or EN ≤ 3 at the end of titration
Evaluate antalgic efficacy criteria | 30 minutes after the initiation of the titration
  Number of patients with EVA ≤ 30 or EN ≤ 3 at 30 minutes
Evaluate antalgic efficacy criteria | From the beginning of the titration until the end of the titration- assessed up to one day
  Number of patients treated only by exclusive inhalation titration with EVA ≤ 30 or EN ≤ 3
Evaluate antalgic efficacy criteria | From the beginning of the titration until the end of the titration- assessed up to one day
  Quantity of of co-analgesia administered from the beginning of the titration
Evaluate antalgic efficacy criteria | 1hour after the initiation of the titration
  Number of patients with EVA ≤ 30 or EN ≤ 3 after 60 minutes
Evaluate antalgic efficacy criteria | 2hours after the initiation of the titration
  Number of patients with EVA ≤ 30 or EN ≤ 3 after 120 minutes
Assess the feasibility of an aerosol titration (compliance to the protocol) | From the beginning of the titration until the end of the aerosol titration- within one hour after the start of the titration
  Number of deviations from protocol
Safety-Proportion of Sleepy patients (Ramsay score = 3) (adverse events) | Until 3hours after the end of the titration
  Proportion of Sleepy patients (Ramsay score = 3)
Safety- incidence of minor side effects in each arm of which neurovegetative usually known and related to opiates (nausea, vomiting, urine retention, ...) | Until 3hours after the end of the titration
  incidence of minor side effects in each arm of which neurovegetative usually known and related to opiates (nausea, vomiting, urine retention,
  ...)
Safety- Proportion of serious adverse events in each arm | Until 3hours after the end of the titration
  Proportion of serious adverse events in each arm

CONTACTS AND LOCATIONS:
Locations (20):
- France (20):
  - CH Agen-Nérac, Agen
  - CHI Robert Ballanger, Aulnay-sous-Bois
  - AP-HP, Bobigny
  - CHU Hôpitaux BORDEAUX, Bordeaux
  - CHU de Caen, Caen
  - CHU Gabriel Montpied, Clermont-Ferrand
  - CH Eure Seine Hôpital d'Evreux, Évreux
  - CHU Grenoble, Grenoble
  - GH Le Havre, Le Havre
  - CH Le Mans, Le Mans
  - CHRU de Lille, Lille
  - Hospices civils de Lyon, Lyon
  - CHU Nice, Nice
  - Hopital COCHIN, Paris
  - Hôpital Lariboisière, Paris
  - La Pitié Salpétrière, Paris
  - CHU-Hôpitaux de Rouen, Rouen
  - Hôpital Bichat-Claude Bernard, Saint-Ouen
  - Chu Strasbourg, Strasbourg
  - chu de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lvovschi VE, Joly J, Lemaire N, Maignan M, Canavaggio P, Leroi AM, Tavolacci MP, Joly LM. Nebulized versus intravenous morphine titration for the initial treatment of severe acute pain in the emergency department: study protocol for a multicenter, prospective randomized and controlled trial, CLIN-AEROMORPH. Trials. 2019 Apr 11;20(1):209. doi: 10.1186/s13063-019-3326-3. PMID 30975187